CLINICAL TRIAL: NCT06104137
Title: MOOC Applications Related to Shared Decision Making in Bariatric Surgery
Acronym: MARS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: South Tyneside and Sunderland NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 322726
Record Dates: First submitted 2023-04-18; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Bariatric Surgery Candidate; Shared Decision Making; Informed Consent
MeSH Terms: interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: double blinded RCT The study design is a randomised clinical trial with two arms. The trial will be double blinded to the consultant surgeon seeing them in clinic and to the assessor of recall but not blinded to the patient. Power calculations showed that to detect an improvement of 20% in the primary outcome measure of recall in the experiment group, with a two-sided 5% significance level and a power of 80% and a drop out rate of 10%, a sample size of 40 patients per arm is necessary.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomisation Method and Blinding Patients who are eligible and consented to participate in the study will be randomised to either the trial group or the control group with use of the sealed envelope method. The randomization will be blocked with use of random permuted blocks in groups of two, four, or six to help ensure that the groups are balanced. A piece of paper that has the phrase "MOOC" or "Control" will be placed in- side an envelope. MOOC patients will have the login and password in the envelope for access.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MOOC group (Experimental): If a patient chooses to take part and is randomly allocated to the MOOC group, a member of research team will issue them with details of how to access the course. Three to six weeks later the research team will contact them to test their recall over the phone of some important information about bariatric surgery. At six week's after the procedure, the research team will send them a copy of the SDM Q9 questionnaire to complete and send back. This is a questionnaire that asks about satisfaction with the shared decision making process.
  Interventions: Other: course (MOOC) patient education
- non MOOC group (Active Comparator): If a patient is randomly allocated to the non MOOC group, they will also receive a recall test and a questionnaire after the consultant appointment in order to compare the two groups.
  Interventions: Other: standard patient consent process

INTERVENTIONS:
Other: course (MOOC) patient education — this is a massive open online course created by us for patient education. Patients will be given a login and password to access the MOOC from their own computer. The MOOC has 3.5 hours of content and patients will be given 3 weeks to complete.
  Arms: MOOC group
Other: standard patient consent process — standard consenting and shared decision making in the clinic
  Arms: non MOOC group

SUMMARY:
What is this trial ? A major aim in surgery is to consent patients appropriately for procedures. This is known as shared decision making. It is the clinician's duty to provide patients with the information they need to weigh up the risks and benefits of surgery and come to an informed decision. The investigators have created a patient information course on bariatric surgery on a platform known as a Massive Open Online Course (MOOC). This platform will host the course and will involve videos, written material and a number of questions to test the patient's understanding. The course will be undertaken after patients have completed Tier 3 and been discussed at the Tier 4 MDT (multidisciplinary team) and before the first consultant appointment to discuss surgical options.

If patients choose to participate, they will be randomly allocated to either undertake the patient information course or not to undertake the course and just undergo the standard consenting process.

The actual timeline of the bariatric journey will be unaffected by participation in the trial. The consultant will not know of patient participation and patients will be asked not to disclose it.

What is involved? The patients will have been invited by one of the researchers, via a telephone call, and they will have sent the patient information for them to read.

Their appointments and schedule will remain the same in spite of participation. If they choose to take part and are randomly allocated to the MOOC group, a member of research team will issue them with details of how to access the course. Three to six weeks later the research team will contact them to test their recall over the phone of some important information about bariatric surgery. At six week's after the procedure, the research team will send a copy of the SDM Q9 (shared decision making Q9) questionnaire to complete and send back. This is a questionnaire that asks about satisfaction with the shared decision making process. If a patient is randomly allocated to the non MOOC group, they will also receive a recall test and a questionnaire after the consultant appointment in order to compare the two groups.

What is the purpose of the trial? The purpose of this study is to find out if using a patient information course on a massive open online course platform (MOOC) is useful to help the consent process by testing patient recall and also to test satisfaction with the shared decision making process compared to what current practice is.

DETAILED DESCRIPTION:
The consenting process is not merely signing a form to allow an intervention or procedure to happen but is a process that allows the sharing of information regarding the procedure which concerns it's benefits, risks and alternatives.

Shared decision making can therefore be defined as a two way process that allows patients to express their preferences and opinions regarding pros, cons and alternatives to a particular procedure and allows the clinician to explain these pros, cons and alternatives on an individual basis. The Royal College of Surgeons has produced guidelines on shared decision making and consent, highlighting the paradigm shift that has occurred in the last ten years in this regard from what was traditionally a more paternalistic unidirectional approach. The College guidelines go further in recommending clinicians to encourage patients to seek web based and other information.

Despite this and the favourable view of both clinicians and patients towards shared decision making, it is clear that it is still in its infancy as highlighted in a 2018 systematic review by de Mik et al. This systematic review of thirty two studies highlights a need for further research with regards to interventions to improve shared decision making. Moreover, reviews from the NHS litigation authority claims against 11 surgical specialties over a ten year period revealed that failure to adequately consent was one of the three leading causes of claim with an estimated £1.5 billion paid out to claimants from 2004 to 2014. It is in the clinician's and patient's benefit for the decision making process to be robust and adequate. It is clear the shared decision making process needs to evolve in practice and where researchers of this study feel Massive Open Online Courses (MOOCs) can play a role.

Massive Open Online Courses have existed as a disruptor in the education sector and allow short courses to a large unrestricted and undifferentiated number of students, on a flexible basis on a wide variety of subjects. Courses are considered more democratic and accessible than traditional higher education courses as they are more inclusive, largely have no pre-requisites and usually free of charge from a range of higher education institutions. MOOCs can also reduce the need for human capital, allow for templates for creation of further courses/patient decision aids and reduce costs of information dissemination. They are also more sustainable and interactive than traditional patient leaflets, can be updated easily and usually involve small tests and certificates as proof of completion as well as being more environmentally friendly.

Thus the trial aims to cover two main unexplored concepts. The first is the feasibility of engaging patients and clinicians in MOOC creation for bariatric surgery. The second is trialing the MOOC in terms of utility as a patient decision aid versus traditional methods of patient information dissemination, which in the researcher's case is a patient leaflet and traditional consenting process. Utility would be investigated by means of ability to recall information and also patient satisfaction with the process using a validated questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age and over who are able to read and write
* Patients who are eligible for tier 4 bariatric services having completed a Tier 3 weight loss programme which is standard criteria for eligibility to have bariatric surgery.

Exclusion Criteria:

* Patients without access to smartphone or a computer are also excluded
* Patients who are having revisional bariatric surgery
* Patients must also have a suitable grasp of the English language in order to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2025-08-04 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
recall testing | 3-6 weeks after recruitment
  a mark out of ten for blinded recall testing by a questionnaire asked of all patients in the trial. Zero is the minimum and the maximum reached is 10.

SECONDARY OUTCOMES:
satisfaction with shared decision making process | 6 weeks post operatively
  validated SDM Q9 questionnaire, marked from 0 to 45, 45 being highest possible score and 0 being the lowest. Higher score indicates higher satisfaction with shared decision making process.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: this is the MOOC the team have created in a prototype form — https://marsbartrialstsft.thinkific.com/courses/bariatric-surgery-for-patients

DOCUMENTS (1):
  • Study Protocol (2023-08-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT06104137/Prot_000.pdf